CLINICAL TRIAL: NCT01574950
Title: The Impact of Impaired Cerebral Autoregulation on the Development of Postoperative Delirium in Elderly Patients Undergoing Spine Surgery
Brief Title: Impact of Impaired Cerebral Autoregulation on Postoperative Delirium in Elderly Patients Undergoing Spine Surgery
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Charles Brown, MD, Principal Investigator, Johns Hopkins University
Other Study IDs: NA_00051796
Record Dates: First submitted 2012-02-16; First posted 2012-04-10 (Estimated); Last update posted 2015-10-26 (Estimated); Status verified 2015-10

CONDITIONS: Delirium
Keywords: Delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No

SUMMARY:
Delirium (confusion) after surgery is common and associated with a longer hospitl stay and increased hopsital cost. There is very little information available about how often delirium occurs and the complications associated with it. Elderly patients are at high risk for delirium after surgery. This research is being done to measure how often delirium after spine surgery occurs and to see if there are ways to predict if delirium will develop. The results from this study will provide important information on a possible mechanism and predictor of delirium.

DETAILED DESCRIPTION:
Delirium (confusion) after surgery is common and associated with a longer hospitl stay and increased hopsital cost. This research is being done to measure how often delirium after spine surgery occurs and to see if there are ways to predict if delirium will develop. We hypothesize that impaired cerebral autoregulation may be a possible mechanism for postoperative delirium. We will measure intraoperative cerebral autoregulation and assess the relationship with postoperative dleirium. The results from this study will provide important information on a possible mechanism and predictor of delirium.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 70 years old,
2. Undergoing any lumbar spine surgery, posterior cervical spine surgery, or anterior cervical spine surgery > 2 levels

Exclusion Criteria:

1. MMSE < 15
2. Delirium at baseline
3. Inability to speak and understand English
4. Severe hearing impairment, resulting in inability to converse.
5. Planned use of intraoperative ketamine
6. Planned use of intraoperative remifentanil, except for airway management pre-incision.
7. Arterial catheter not planned to be inserted

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population is male and female subjects age 70 years and older that are having spine surgery.
Sampling Method: Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2012-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Incidence of post-operative delirium in elderly patients undergoing spine surgery at Johns Hopkins Hospital | 24 months

SECONDARY OUTCOMES:
Severity of postoperative delirium, using Delirium Rating Scale-Revised-1998, in elderly patients undergoing spine surgery. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Charles Brown, MD, Principal Investigator — The Johns Hopkins University
Locations (1):
- The Johns Hopkins University, Baltimore, Maryland, United States